CLINICAL TRIAL: NCT03948945
Title: Efficacy and Safety of Profile HaloTM Dual-wavelength Fusion Fractional Laser on the Treatment of Facial and Neck Photoaging: a Self-controlled Trial.
Brief Title: Efficacy and Safety of Profile HaloTM Mixed Fractional Laser on Treating of Facial and Neck Photoaging.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: xjpfW (Other)
Collaborators: Air Force General Hospital of the PLA (Other Government); First Hospital of China Medical University (Other); Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, xjpfW, Head of Dermatology, Xijing Hospital
Organization: Xijing Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: XijingH-PF-20150705
Record Dates: First submitted 2019-05-10; First posted 2019-05-14 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Photoaging
Keywords: Fractional Laser; Photoaging; Treatment; Halo

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- before treatment (No Intervention): The patient with facial and neck photoaging did not receive laser treatment.
- after treatment (Experimental): The patient with facial and neck photoaging received Profile HaloTM mixed fractional laser treatment
  Interventions: Radiation: Profile HaloTM Mixed Fractional Laser

INTERVENTIONS:
Radiation: Profile HaloTM Mixed Fractional Laser — Profile HaloTM fractional laser is the world's first hand tool with nonablative and ablative fractional laser. It includes a nonablative fractional laser with a wavelength of 1470 nm and an ablative fractional laser with a wavelength of 2940 nm. It has a good therapeutic effect on skin aging.
  Arms: after treatment

SUMMARY:
1. Fractional laser has become an important laser modality in management of a number of skin conditions and photoaging. Fractional photothermolysis is the fractional emission of light into microscopic treatment zones, creating small columns of injury to the skin in a pixilated fashion. Epidermal and dermal disruptions occur in these focal zones of thermal injury, stimulating dermal collagen production and elastic tissue formation. Fractional laser has been used successfully to treat photodamage and overall dyschromia in the Caucasian population. However, there is not much improvement in Asian population.
2. Photoaging refers to the skin caused by intense and chronic exposure to sunlight. The visible effects of photoaging are fine wrinkles, mottling, pigmentation and roughness of the skin. These changes are usually associated with chronologic aging. However, photoaging is not a good indicator of chronologic age. It just makes a person look older than his or her chronologic age. Skin ageing may be divided into two processes: intrinsic ageing and extrinsic ageing (or photoageing). Both are accompanied by changes in the morphological and biomechanical properties of skin.
3. Profile HaloTM dual-wavelength fusion fractional laser is the first hand tool in the world that integrates ablative and non-ablative fractional lasers. It includes a non-ablative fractional laser with a wavelength of 1470nm and an ablative fractional laser with a wavelength of 2940nm. A day after treatment, new epithelial tissue began to appear, and the necrotic epidermis formed microepidermal necrotic debris (MENDs). MENDs were surrounded by keratin 2-7 days after treatment, and collagen sequence in MTZs was changed 7 days later. The 2940 ablative fractional laser can be added with 20-100 micron lattice stripping, ensuring safety while enabling MENDs to be peeled off 2 days earlier and reducing the risk of side effects. This makes the laser safe and effective compared with the single fractional laser and reduces the downtime.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be clinically diagnosed by the investigator to facial photoaging dover 2-4 and cervical stripe Fitzpatrick 1-2.5
* no other treatment was performed for the skin lesions for half a year before the treatment
* patients with a "no" in any of the above criteria are not eligible for inclusion

Exclusion Criteria:

* subjects with a recent history of exposure to sunlight;
* subjects allergic to topical anesthesia;
* subjects with scar constitution;
* subjects with skin malignant tumors or precancerous lesions; .subjects with diabetes, heart disease, epilepsy, connective tissue disease, etc.
* subjects who Pregnant or breast feeding;
* subjects with recent skin infections (such as viruses, bacteria, etc.);
* ther methods are being used to treat subjects with similar diseases;
* subject who have taken isotretinoin A in the past year; .subject with facial dermatitis.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
VISIA skin test | change from week0 to week48
  With fast capture times and lighting modes designed to enhance the visualization of skin features, VISIA®-CR (Canfield Scientific, Inc. USA) is the standard in repeatable clinical imaging. Visia CR imaging system can be used to assess the skin wrinkles, texture, pores and elasticity

SECONDARY OUTCOMES:
Neck (Fitzpatrick wrinkle grading) | week0,week48
  Level 0: no wrinkles, no visible wrinkles and continuous skin lines; Level 0.5: very shallow wrinkles visible to the naked eye Level 1: fine wrinkles, slight depressions visible to naked eye Level 1.5: visible wrinkles and clear depressions with a depth of <0.01mm; Level 2: medium wrinkles. It can be clearly seen that the depth of wrinkles is 1-2mm.
  Level 2.5: obvious visible wrinkles with a depth of 2-3mm; Level 3: deep wrinkles, visible deep marks, depth greater than > 3mm
Glogau Classification of Photoaging | change from week0 to week48
  I： Mild 28-35 years old No wrinkles Early Photoaging: mild pigment changes, no keratosis, minimal wrinkles, minimal or no makeup； II： Moderate 35-50 years old Wrinkles in motion Early to Moderate Photoaging: Early brown spots visible, keratosis palpable but not visible, parallel smile lines begin to appear, wears some foundation； III： Advanced 50-65 years old Wrinkles at rest Advanced Photoaging: Obvious discolorations, visible capillaries (telangiectasias), visible keratosis, wears heavier foundation always； IV： Severe 60-75 years old Only wrinkles Severe Photoaging: Yellow-gray skin color, prior skin malignancies, wrinkles throughout-no normal skin, cannot wear makeup because it cakes and cracks

CONTACTS AND LOCATIONS:
Overall Officials: Gang Wang, Prof, Principal Investigator — Dermatology Derpartment of Xijing Hospital

IPD SHARING:
Plan to Share IPD: No